CLINICAL TRIAL: NCT06079489
Title: The Effect of Telerehabilitation-Based Structured Exercise Program in Video Game-Addicted Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: buhucgun03
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Video Game Addiction
MeSH Terms: conditions — Technology Addiction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants were advised to repeat the brochure-based exercises 3 days a week for 8 weeks. Correct sitting and standing positions and ergonomic materials were also explained in detail. Participants' adherence to the exercise program was tracked by an exercise diary.
  Interventions: Other: Brochure-Based Exercise Program
- Experimental Group (Experimental): Progressive physical fitness and posture exercises were given via telerehabilitation 3 days a week for 8 weeks. Specific exercises for upper extremities, lower extremities, neck, trunk and lower back were selected and progressed by changing the frequency, duration and variety within the program. All exercises were performed under the supervision of a physiotherapist during video conference calls lasting an average of 40 minutes. Correct sitting and standing positions and ergonomic materials were also explained in detail. Participants' adherence to the exercise program was tracked by an exercise diary.
  Interventions: Other: Telerehabilitation-Based Structured Exercise Program

INTERVENTIONS:
Other: Brochure-Based Exercise Program — Simple posture exercises
  Arms: Control Group
Other: Telerehabilitation-Based Structured Exercise Program — Progressive physical fitness and posture exercises
  Arms: Experimental Group

SUMMARY:
The increasing use of computers and mobile devices due to advancing technology has brought with it some negative consequences such as video game addiction. Research has shown that playing video games for too long can lead to a number of acute and chronic serious musculoskeletal problems that can negatively affect health. The aim of the present study is to investigate the effect of telerehabilitation-based structured exercise program in video game-addicted adults and compare these effects with the effect of brochure-based exercise. Postural assessments, pain assessments, fine motor skill assessments, grip strength measurements, and reaction time assessments were performed. All assessments were repeated before and after the 8-week program for both groups. Participants in the EG were given a telerehabilitation-based structured exercise program for an average of 40 minutes three days a week for 8 weeks. Participants in the CG were given brochure-based exercises three days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-40 years old
* Having a score of ≥30 on the Game Addiction Inventory for Adults (GAIA)
* Volunteering to participate in the study
* Having high-speed internet, a camera, and a microphone

Exclusion Criteria:

* Having a neurological/orthopedic condition that would prevent exercise
* Having a cognitive impairment
* Having a vision or hearing loss

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Assessment | 1-2 minutes
  The pain was assessed with the 10-cm VAS. The participants used the VAS to make an assessment of their own pain, with 0 representing no pain, and 10 cm representing severe pain.
Fine Motor Skill Assessment | 4-5 minutes
  The fine motor skill was assessed with the 9-Hole Peg Test. It is a simple, fast test that requires minimal space and equipment and evaluates fine upper motor function. In this test, the patient is asked to insert the pegs into the holes in the desired order and collect them back. The duration of the test is measured by a specialist via a stopwatch.
Posture Assessment | 5-10 minutes
  Posture was assessed with the PostureZone Posture Application. The PostureZone mobile application, which can be downloaded free of charge on both Android and iOS via smartphone, will be used to evaluate the static postures of the participants. It is an application developed for clinicians that assess static posture. The participant is photographed with minimal clothing on, certain pivot points are marked, and the deviations of these points relative to the vertical-horizontal planes are determined.
Hand Reaction Assessment | 10-15 minutes
  Hand Reaction was assessed with the Nelson Hand Reaction Test. The participant sits on a chair with his forearm and hand in a comfortable position on the table. The tester holds the end of the ruler. The participant is asked to catch the ruler. Twenty rials are performed. The lowest 5 and highest 5 attempts are discarded and the average of the remaining 10 attempts is recorded as the result.
Handgrip Strength Assessment | 4-5 minutes
  Jamar Hydraulic Hand Dynanometer was used to assess handgrip strength. Each trial was repeated three times and the average was recorded in kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No